CLINICAL TRIAL: NCT00832390
Title: Study to Assess the Efficacy and Safety of Sitagliptin in Recently Diagnosed, Naive Type 2 Diabetics With Inadequate Glycemic Control on Diet and Exercise
Brief Title: Study to Assess the Efficacy and Safety of Sitagliptin in Recently Diagnosed, Naive Type 2 Diabetics With Inadequate Glycemic Control on Diet and Exercise (0431-158)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431-158; 2009_525
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Results first posted 2009-07-31 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): sitagliptin
  Interventions: Drug: sitagliptin phosphate

INTERVENTIONS:
Drug: sitagliptin phosphate — Patients will receive sitagliptin with metformin for 24 weeks, given as oral tablets
  Other Names: MK0431

SUMMARY:
After 24 weeks of treatment evaluate the efficacy and security.

ELIGIBILITY:
Inclusion Criteria:

* Patients Being Treated With Metformin
* Patients With Hba1c Between 6.5 % And 12.0%.
* Type 2 DM

Ages: 30 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-02-14 (Actual); Primary Completion 2008-07-11 (Actual); Study Completion 2008-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single site study with patients recruited in Principal Investigator's private practice, Mexico City.
  First Patient In: 14Feb2007. Last Patient's Last Visit: 11Jul2008
Pre-assignment Details: Treatment naïve patients (30 to 78 years of age) with inadequate glycemic control on diet/exercise were assigned to treatment with sitagliptin alone (A1C 6.5 to <8%), sitagliptin + metformin as initial combination therapy (A1C 8-12%), or standard care.
Groups:
- Standard Care Regimen: Patients in the "standard care" group were to receive usual care per practice but not to be treated with sitagliptin or another DPP-4 inhibitor. As prespecified in the protocol, no efficacy was to be assessed in this group.
Period: Overall Study
Arm/Group | Sitagliptin 100 mg q.d. (Once Daily) | Sitagliptin 100 mg q.d. (Once Daily) and Metformin | Standard Care Regimen
Started | 12 | 16 | 1
Completed | 12 | 16 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg q.d. (Once Daily) | Sitagliptin 100 mg q.d. (Once Daily) and Metformin | Standard Care Regimen | Total
Number analyzed (Participants) | 12 | 16 | 1 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (14.1) | 52.5 (9.3) | 51.0 (0.0) | 54.62 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 1 | 20
  Male | 6 | 3 | 0 | 9
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.4 (10.0) | 28.9 (5.2) | 26.0 (0.0) | 28.14 (7.41)
Glycosylated Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent] | 7.1 (0.6) | 8.6 (1.4) | 6.9 (0.0) | 7.96 (1.33)
Time Since Diagnosis of Diabetes [Mean (Standard Deviation); unit: Years] | 5.3 (7.0) | 6.2 (6.0) | 5.2 (0.0) | 5.82 (6.25)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 24
Description: Week 24 A1C minus baseline (Week 0) A1C. The unit for A1C is "percent". Thus, this measure represents a difference of percent values.
Time Frame: Baseline and 24 Weeks
Measure: Mean (95% Confidence Interval); unit: Percent Difference
Arm/Group | Sitagliptin 100 mg q.d. (Once Daily) | Sitagliptin 100 mg q.d. (Once Daily) and Metformin | Standard Care Regimen
Number analyzed (Participants) | 12 | 16 | 1
Percent Difference | -0.2 [-0.9 to 0.5] | -1.0 [-2.1 to -0.1] | 0.0 [0.0 to 0.0]

ADVERSE EVENTS:
Arm/Group | Sitagliptin 100 mg q.d. (Once Daily) | Sitagliptin 100 mg q.d. (Once Daily) and Metformin | Standard Care Regimen
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/16 | 0/1
Other Adverse Events (participants affected / at risk) | 1/12 | 0/16 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg q.d. (Once Daily) (N=12) | Sitagliptin 100 mg q.d. (Once Daily) and Metformin (N=16) | Standard Care Regimen (N=1)
Hypertension (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Few participants were recruited into this single-site study as the investigator preferred the use of initial combination therapy.

Protocol deviations may have occurred that resulted in quality issues associated with reporting of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.